CLINICAL TRIAL: NCT01534468
Title: Evaluation of Priming by Pandemic Live Attenuated Influenza Vaccine (LAIV) on the Subsequent Response to Inactivated H7N7 Vaccine in Healthy Adults: A Non-Randomized, Open Label Study
Brief Title: Evaluating the Safety and Immune Response of an H7N7 Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: URMC 11-001
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Influenza A Subtype H7N7 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Previous H7N7 ca LAIV recipients (Experimental): Participants in Group 1 will have previously received an H7N7 ca LAIV. In this study, they will receive one intramuscular (IM) injection of the H7N7 vaccine at study entry.
  Interventions: Biological: Monovalent Influenza Subvirion Vaccine, H7N7
- Group 2: Previous H7N3 ca LAIV recipients (Experimental): Participants in Group 2 will have previously received an H7N3 ca LAIV. In this study, they will receive one IM injection of the H7N7 vaccine at study entry.
  Interventions: Biological: Monovalent Influenza Subvirion Vaccine, H7N7
- Group 3: Previous H2N3 ca LAIV recipients (Experimental): Participants in Group 3 will have previously received an H2N3 ca LAIV. In this study, they will receive one IM injection of the H7N7 vaccine at study entry.
  Interventions: Biological: Monovalent Influenza Subvirion Vaccine, H7N7
- Group 4: Vaccine-naive participants (Experimental): Participants in Group 4 will have not previously received a LAIV. In this study, they will receive one IM injection of the H7N7 vaccine at study entry.
  Interventions: Biological: Monovalent Influenza Subvirion Vaccine, H7N7

INTERVENTIONS:
Biological: Monovalent Influenza Subvirion Vaccine, H7N7 — At study entry, all participants will receive one IM injection of approximately 45 micrograms of inactivated Monovalent Influenza Subvirion Vaccine, H7N7.

SUMMARY:
H7N7 is one type of influenza virus that may pose a threat to humans if an outbreak occurs. This study will evaluate the safety and immune response to an H7N7 vaccine in people who have previously received a live attenuated influenza vaccine (LAIV) as part of a research study and people who have not previously received a LAIV.

DETAILED DESCRIPTION:
Influenza A viruses are widely found in nature and can infect a wide variety of birds and mammals, including humans. Some types of influenza A viruses are more likely to spread from animals to humans, and researchers are interested in monitoring these viruses and developing potential vaccines for them. H7N7 is one type of influenza A virus. In recent years, there have been several H7N7 outbreaks among humans, and the development of an H7N7 vaccine is a high priority. This study will enroll two groups of participants: people who have previously received one of three types of a pandemic LAIV as part of a research study and people who have not previously received a LAIV vaccine. The purpose of this study is to evaluate the safety and immunogenicity of a single dose of an inactivated H7N7 vaccine in these two groups of participants.

At a baseline study visit, all participants will undergo a medical history review, physical examination, vital sign measurements, blood collection, and nasal secretion collection. Female participants will provide a urine sample for pregnancy testing. All participants will then receive one intramuscular (IM) injection of the H7N7 study vaccine in their upper arm. They will remain in the clinic for 30 minutes for observation and monitoring. Participants will monitor and record any adverse symptoms between study visits. Additional study visits will occur at Days 4, 7, 14, 28, 56, and 180. At select study visits, participants will undergo a medical history review, physical examination, and nasal secretion collection. Blood collection will occur at each visit; some blood samples may be stored for future research.

ELIGIBILITY:
Inclusion Criteria:

* Previous participant in a study of pandemic LAIV or H7-naive participant, as described in the protocol
* Adult males and non-pregnant females between 18 and 50 years of age
* In good general health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator
* Agree to storage of blood specimens for future research
* Available for the duration of the trial
* Willing to participate in the study as evidenced by signing the informed consent document
* Female participants must agree to use effective birth control methods for the duration of the study. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Pregnant, as determined by a positive beta-human chorionic gonadotropin (HCG) test
* Currently breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies, including urine testing. Alanine transaminase (ALT) levels more than twice the upper limit of normal, or otherwise clinically significant as determined by the principal investigator (PI), will be exclusionary at baseline, prior to vaccination.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
* Previous enrollment in an inactivated H7N7 influenza vaccine trial
* Seropositive to the H7N7 influenza A virus (serum HAI titer greater than 1:8) for H7-naive participants
* Positive urine drug toxicity test indicating use of drugs of abuse
* Medical, occupational, or family problems as a result of alcohol or illicit drug use in the 12 months prior to study entry
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* History of anaphylaxis
* History of Guillain-Barre syndrome
* Positive ELISA and confirmatory Western blot tests for HIV-1
* Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay [RIBA]) for hepatitis C virus (HCV)
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination
* History of a surgical splenectomy
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination
* Travel to the Southern Hemisphere within 14 days prior to study vaccination
* Travel on a cruise ship within 14 days prior to study vaccination
* Current involvement with the poultry industry, i.e., direct contact with poultry within the 14 days prior to study entry or after the study completion
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination
* Allergy to eggs or egg products

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events that occur during the acute monitoring phase of the study | Measured through Day 7
Development of serum antibody assessed by either hemagglutination inhibition (HAI) or micronucleus (MN) assays | Measured through Day 180

SECONDARY OUTCOMES:
Development of a significant increase in nasal secretion hemagglutinin (HA)-specific antibody, as assessed by enzyme-linked immunosorbent assay (ELISA) | Measured through Day 180
Development of greater than 200 influenza-specific interferon-gamma (IFN-γ)-secreting cells per million lymphocytes, as assessed by enzyme-linked immunosorbent spot (ELISPOT) | Measured on Day 28
Detection of influenza-specific immunoglobulin G (IgG)- or immunoglobulin A (IgA)-secreting B cells, as assessed by antibody secreting cells (ASC) assay | Measured on Day 7

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Halliley JL, Khurana S, Krammer F, Fitzgerald T, Coyle EM, Chung KY, Baker SF, Yang H, Martinez-Sobrido L, Treanor JJ, Subbarao K, Golding H, Topham DJ, Sangster MY. High-Affinity H7 Head and Stalk Domain-Specific Antibody Responses to an Inactivated Influenza H7N7 Vaccine After Priming With Live Attenuated Influenza Vaccine. J Infect Dis. 2015 Oct 15;212(8):1270-8. doi: 10.1093/infdis/jiv210. Epub 2015 Apr 2. PMID 25838266
- [Derived] Babu TM, Levine M, Fitzgerald T, Luke C, Sangster MY, Jin H, Topham D, Katz J, Treanor J, Subbarao K. Live attenuated H7N7 influenza vaccine primes for a vigorous antibody response to inactivated H7N7 influenza vaccine. Vaccine. 2014 Nov 28;32(50):6798-804. doi: 10.1016/j.vaccine.2014.09.070. Epub 2014 Oct 16. PMID 25446831